CLINICAL TRIAL: NCT07295535
Title: Analysis of the Specificity and Persistence of Nasal Immune Responses to Respiratory Viral Antigens in Immunocompromised and Healthy Cohorts
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefania Mantovani, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Nasal Immunity Study
Record Dates: First submitted 2025-12-01; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Immuno-modulation; Immuno-suppression; Immunocompromised Patients; Healthy Subjects; Oncological Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal Swabs, Isolated PBMCs and Serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompromised patients: Participants with medical conditions or treatments associated with significant impairment of the immune system. This may include organ or stem cell transplants, ongoing immunosuppressive therapies, documented genetic immunosuppression.
- Healthy Volunteers: No underlying medical conditions declared, no clinical history of immunodeficiency or use of immunosuppressive medications.

SUMMARY:
The goal of this observational study is to characterize nasal mucosal immunity to respiratory viruses, such as SARS-CoV-2, in immunocompromised individuals and healthy volunteers.

The study involves adults of any sex, between 18 and 90 years old, including both immunocompromised patients with medical conditions or treatments that can affect immune cell functions and healthy controls with no underlying medical conditions declared, no clinical history of immunodeficiency or use of immunosuppressive medications.

Researchers will compare immunocompromised participants to healthy volunteers to determine how underlying immunodeficiency and related treatments affect immune cell composition and virus-specific responses.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Participants must have signed an informed consent form.
* Age Range: Participants aged between 18 and 90 years.
* Healthy Immunocompetent Donors: no underlying medical conditions declared, no clinical history of immunodeficiency or use of immunosuppressive medications.
* Immunocompromised Patients: subjects with medical conditions or treatments associated with significant impairment of the immune system. This may include organ or stem cell transplants, ongoing immunosuppressive therapies, documented genetic immunosuppression.

Exclusion Criteria:

* Pregnant or lactating women.
* Individuals unable to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will take place at primary care clinic. Immunocompromised participants will be selected based on their regular visits, while healthy donors will be recruited through hospital and research networks.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-27 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of cytokines produced by viral-specific nasal and peripheral T cells. | Assessed at 4 periodic intervals, approximately 45 days apart, based on clinical follow-up visits, starting from the beginning of enrollment up to 6 months.

SECONDARY OUTCOMES:
Phenotypic characterisation of nasal and peripheral immune cells. | Measured at the time of enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No